CLINICAL TRIAL: NCT04734028
Title: Platelet Function and genoType-Related Long-term progGosis in DES-treated Patients : A Consortium From Multi-centered Registries
Brief Title: PTRG-DES Consortium
Acronym: PTRG
Status: Completed | Type: Observational
Sponsor: Gyeongsang National University Hospital (Other)
Collaborators: Korean Society of Interventional Cardiology (Unknown)
Responsible Party: Sponsor
Other Study IDs: PTRG
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease; Clopidogrel, Poor Metabolism of; Platelet Dysfunction; Stent Thrombosis
Keywords: Asian population; VerifyNow assay; Genotype; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PTRG-DES registry: After DES implantation, CAD patients were treated with DAPT with clopidogrel and aspirin. During hospitalization, their platelet function, genotype and inflammation biomarker were evaluated.
  Interventions: Drug: Clopidogrel Tablets

INTERVENTIONS:
Drug: Clopidogrel Tablets — DES-treated patients were treated with clopidogrel 75 mg daily and aspirin 100 mg daily
  Other Names: aspirin

SUMMARY:
The PTRG-DES consortium is a coalition composed of multi-center, real-world registries including CAD patients treated with DES in South Korea. From 9 academic registries in Korea, a total of 13,160 patients were enrolled for this database between July 2003 and August 2018. The aim of the study was to investigate long-term prognostic implications of platelet function and genotypes after DES implantation for significant CAD in South Korea.

DETAILED DESCRIPTION:
The investigators enrolled patients treated with DES during DAPT including clopidogrel who had at least one of VerifyNow test (PRU and ARU) and genotyping. In this consortium, the investigators tried to find the unique characteristics of East Asians based on platelet function, genotype and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients at every centre successfully treated with one or more DES approved by the US FDA or CE mark and who were adequately loaded with clopidogrel were eligible for enrolment, regardless of patient or lesion complexity.

Exclusion Criteria:

* the occurrence of a major complication during the procedure or before platelet function testing, or if bypass surgery was planned after PCI.
* Any P2Y12 inhibitor other than clopidogrel
* PCI strategy other than DES
* Needed oral anticoagulant (e.g. atrial fibrillation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Significant CAD patients treated with uneventful DES implantation
Sampling Method: Non-Probability Sample
Enrollment: 13160 (Actual)
Dates: Start 2003-07-09 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
MACCE | upto 10 years
  All-cause death, MI, stroke or stent thrombosis

SECONDARY OUTCOMES:
Major bleeding | upto 10 years
  BARC type 3-5 bleeding
MACE1 | upto 10 years
  CV death, MI and stent thrombosis
MACE2 | upto 10 years
  CV death, MI, stent thrombosis and revascularization
Each clinical event | upto 10 years
  all-cause death, CV death, MI, stroke, stent thrombosis, revascularization or major bleeding

OTHER OUTCOMES:
Clinical event according to gender | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to age | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to BMI | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to anemia | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to DM | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to CKD | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to disease entity (AMI vs. non-AMI) | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to LV dysfunction (LV EF) | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to complex PCI | upto 10 years
  prognostic implications of PFT, genotype and CRP
Clinical event according to time point post-PCI | upto 10 years
  prognostic implications of PFT, genotype and CRP

CONTACTS AND LOCATIONS:
Overall Officials: Do-Sun Lim, MD, PhD, Study Chair — Korea University Anam Hospital, Korea University School of Medicine
Locations (1):
- Gyeongsang National University Changwon Hospital, Changwon, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
If there are the chances of collaboration work, we will share IPD with other groups.

REFERENCES:
- [Result] Kim HK, Tantry US, Smith SC Jr, Jeong MH, Park SJ, Kim MH, Lim DS, Shin ES, Park DW, Huo Y, Chen SL, Bo Z, Goto S, Kimura T, Yasuda S, Chen WJ, Chan M, Aradi D, Geisler T, Gorog DA, Sibbing D, Lip GYH, Angiolillo DJ, Gurbel PA, Jeong YH. The East Asian Paradox: An Updated Position Statement on the Challenges to the Current Antithrombotic Strategy in Patients with Cardiovascular Disease. Thromb Haemost. 2021 Apr;121(4):422-432. doi: 10.1055/s-0040-1718729. Epub 2020 Nov 10. PMID 33171520
- [Derived] Kang J, Park S, Park KW, Joo HJ, Chang K, Park Y, Song YB, Ahn SG, Suh JW, Lee SY, Cho JR, Her AY, Jeong YH, Kim BK, Kim MH, Shin ES, Lim DS, Hwang D, Han JK, Yang HM, Koo BK, Kim HS; PTRG Investigators. Long-Term Impact of Platelet Reactivity and Clinical Risk on Clinical Outcomes in Patients With Coronary Artery Disease: Analysis of the PTRG-DES Registry. Circ Cardiovasc Interv. 2025 Oct;18(10):e015737. doi: 10.1161/CIRCINTERVENTIONS.125.015737. Epub 2025 Sep 22. PMID 40977391
- [Derived] Ahn H, Chu HW, Her AY, Jeong YH, Kim BK, Joo HJ, Chang K, Park Y, Ahn SG, Lee SY, Cho JR, Kim HS, Kim MH, Lim DS, Shin ES, Suh JW; PTRG-DES Consortium Investigators. Effect of Calcium Channel Blockers on Antiplatelet Activity of Clopidogrel in Patients Undergoing Percutaneous Coronary Intervention: Insights from the PTRG-DES Consortium. J Cardiovasc Pharmacol Ther. 2024 Jan-Dec;29:10742484241298150. doi: 10.1177/10742484241298150. PMID 39552592
- [Derived] Kim JH, Lee SJ, Cha JJ, Park JH, Hong SJ, Ahn TH, Kim BK, Chang K, Park Y, Song YB, Ahn SG, Suh JW, Lee SY, Cho JR, Her AY, Jeong YH, Kim HS, Kim MH, Shin ES, Lim DS; PTRG-DES Consortium Investigators. Prognostic Impact of CYP2C19 Genotypes on Long-Term Clinical Outcomes in Older Patients After Percutaneous Coronary Intervention. J Am Heart Assoc. 2024 May 21;13(10):e032248. doi: 10.1161/JAHA.123.032248. Epub 2024 May 18. PMID 38761068
- [Derived] Won KB, Kim HJ, Cho JH, Lee SY, Her AY, Kim BK, Joo HJ, Park Y, Chang K, Song YB, Ahn SG, Suh JW, Cho JR, Kim HS, Kim MH, Lim DS, Kim SW, Jeong YH, Shin ES. Different association of atherogenic index of plasma with the risk of high platelet reactivity according to the presentation of acute myocardial infarction. Sci Rep. 2024 May 13;14(1):10894. doi: 10.1038/s41598-024-60999-3. PMID 38740817
- [Derived] Jin X, Jeong YH, Lee KM, Yun SC, Kim BK, Joo HJ, Chang K, Park YW, Song YB, Ahn SG, Suh JW, Lee SY, Cho JR, Her AY, Kim HS, Lim DS, Shin ES, Kim MH; PTRG-DES Consortium Investigators. Prognostic Implication of Platelet Reactivity According to Procedural Complexity After PCI: Subanalysis of PTRG-DES Consortium. JACC Asia. 2023 Dec 26;4(3):185-198. doi: 10.1016/j.jacasi.2023.10.011. eCollection 2024 Mar. PMID 38463677
- [Derived] Han D, Kim SH, Shin DG, Kang MK, Choi S, Lee N, Kim BK, Joo HJ, Chang K, Park Y, Song YB, Ahn SG, Suh JW, Lee SY, Her AY, Jeong YH, Kim HS, Kim MH, Lim DS, Shin ES, Cho JR; PTRG Investigator. Prognostic Implication of Platelet Reactivity According to Left Ventricular Systolic Dysfunction Status in Patients Treated With Drug-Eluting Stent Implantation: Analysis of the PTRG-DES Consortium. J Korean Med Sci. 2024 Jan 22;39(3):e27. doi: 10.3346/jkms.2024.39.e27. PMID 38258362
- [Derived] Lim S, Hong SJ, Kim JH, Cha JJ, Joo HJ, Park JH, Yu CW, Kim BK, Chang K, Park Y, Song YB, Ahn SG, Suh JW, Lee SY, Cho JR, Her AY, Jeong YH, Kim HS, Kim MH, Shin ES, Lim DS; PTRG Investigators. High platelet reactivity strongly predicts early stent thrombosis in patients with drug-eluting stent implantation. Sci Rep. 2024 Jan 4;14(1):520. doi: 10.1038/s41598-023-50920-9. PMID 38177178
- [Derived] Jeon KH, Jeong YH, Chae IH, Kim BK, Joo HJ, Chang K, Park Y, Song YB, Ahn SG, Lee SY, Cho JR, Her AY, Kim HS, Kim MH, Lim DS, Shin ES, Suh JW; PTRG-DES Consortium Investigators. Implication of diabetic status on platelet reactivity and clinical outcomes after drug-eluting stent implantation: results from the PTRG-DES consortium. Cardiovasc Diabetol. 2023 Sep 7;22(1):245. doi: 10.1186/s12933-023-01976-4. PMID 37679760
- [Derived] Kim SJ, Her AY, Jeong YH, Kim BK, Joo HJ, Park Y, Chang K, Song YB, Ahn SG, Suh JW, Lee SY, Cho JR, Kim HS, Kim MH, Lim DS, Shin ES; PTRG-DES Consortium Investigators. Sex Differences in Midterm Prognostic Implications of High Platelet Reactivity After Percutaneous Coronary Intervention With Drug-Eluting Stents in East Asian Patients: Results From the PTRG-DES (Platelet Function and Genotype-Related Long-Term Prognosis in Drug-Eluting Stent-Treated Patients With Coronary Artery Disease) Consortium. J Am Heart Assoc. 2023 May 2;12(9):e027804. doi: 10.1161/JAHA.122.027804. Epub 2023 Apr 29. PMID 37119080
- [Derived] Lee SH, Jeong YH, Hong D, Choi KH, Lee JM, Park TK, Yang JH, Hahn JY, Choi SH, Gwon HC, Jeong MH, Kim BK, Joo HJ, Chang K, Park Y, Ahn SG, Suh JW, Lee SY, Cho JR, Her AY, Kim HS, Kim MH, Lim DS, Shin ES, Song YB; PTRG-DES Registry Investigators. Clinical Impact of CYP2C19 Genotype on Clopidogrel-Based Antiplatelet Therapy After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2023 Apr 10;16(7):829-843. doi: 10.1016/j.jcin.2023.01.363. Epub 2023 Mar 8. PMID 37045504
- [Derived] Lee SJ, Cha JJ, Jeong YH, Hong SJ, Ahn CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y, Joo HJ, Chang K, Park Y, Song YB, Ahn SG, Suh JW, Lee SY, Cho JR, Her AY, Kim HS, Kim MH, Shin ES, Lim DS, Kim BK; PTRG Investigators. Platelet Reactivity and Clinical Outcomes After Drug-Eluting Stent Implantation: Results From the PTRG-DES Consortium. JACC Cardiovasc Interv. 2022 Nov 28;15(22):2253-2265. doi: 10.1016/j.jcin.2022.09.007. PMID 36423968
- [Derived] Her AY, Jeong YH, Kim BK, Joo HJ, Chang K, Park Y, Song YB, Ahn SG, Suh JW, Lee SY, Cho JR, Kim HS, Kim MH, Lim DS, Shin ES; PTRG-DES Consortium Investigators. Platelet Function and Genotype after DES Implantation in East Asian Patients: Rationale and Characteristics of the PTRG-DES Consortium. Yonsei Med J. 2022 May;63(5):413-421. doi: 10.3349/ymj.2022.63.5.413. PMID 35512743
- See also: Thrombosis and Haemostasis — https://www.thieme-connect.com/products/ejournals/abstract/10.1055/s-0040-1718729